CLINICAL TRIAL: NCT06232655
Title: Study of Cladribine+Venetoclax After Failure of Venetoclax+Hypomethylating Agent in Monocytic AML
Brief Title: Cladribine Venetoclax in Monocytic AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-0273.cc
Record Dates: First submitted 2024-01-19; First posted 2024-01-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Cladribine; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cladribine plus Venetoclax (Experimental): Subjects will receive cladribine at a dose of 5mg/m2 daily via intravenous infusion on days 1 through 5 of a 28 day cycle. Concomitantly, venetoclax will be administered orally at a dose of 100mg on day 1, 200mg on day 2, and 400mg daily on days 3 through 28.
  Interventions: Drug: Cladribine; Drug: Venetoclax
- Alternating Aza/Ven and Clad/Ven (Experimental): Alternating 28-day consolidation cycles of Aza/Ven (even cycles) and Clad/Ven (odd cycles), while those who do not respond will come off the study.
  Interventions: Drug: Cladribine; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Cladribine — A medication used to treat hairy cell leukemia (leukemic reticuloendotheliosis) and B-cell chronic lymphocytic leukemia. Cladribine, sold under the brand name Mavenclad, is used for the treatment of adults with highly active forms of relapsing-remitting multiple sclerosis.
  Other Names: Mavenclad; Leustatin
Drug: Venetoclax — A medication used to treat adults with chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or acute myeloid leukemia (AML).
  Other Names: Venclyxto
Drug: Azacitidine — Medication used for the treatment of myelodysplastic syndrome, myeloid leukemia, and juvenile myelomonocytic leukemia. It is a chemical analog of cytidine, a nucleoside in DNA and RNA.. Azacitidine and its deoxy derivative, decitabine were first synthesized in Czechoslovakia as potential chemotherapeutic agents for cancer.
  Other Names: Vidaza; Onureg
  Arms: Alternating Aza/Ven and Clad/Ven

SUMMARY:
Investigation of Relapsed or refractory AML with a monocytic phenotype after failure of hypomethylating agent+venetoclax

DETAILED DESCRIPTION:
This is an investigator-initiated, open label, single institution, Study to assess the efficacy of Clad/Ven following failure of HMA/Ven in AML with a monocytic phenotype. In cycle 1, subjects will receive cladribine at a dose of 5mg/m2 daily via intravenous infusion on days 1 through 5 and venetoclax 400mg daily (following standard dose escalation over the first 3 days) on days 1 through 28 of a 28 day cycle. A bone marrow biopsy will be performed to assess response on day 28 of cycle 1. Subjects who respond to cycle 1, defined as achieving a CR, CRi, MLFS, or PR per ELN criteria, or a blast reduction of at least 50% from baseline, may continue on alternating 28-day consolidation cycles of Aza/Ven (even cycles) and Clad/Ven (odd cycles). Cycles will continue unless the subject needs to be removed from the study due to disease progression, treatment failure (defined as failure to achieve CR, CRi, or MLFS after 4 cycles of treatment), intolerance or toxicity, patient preference, or other reasons.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if they meet the following criteria within 28 days prior to the first day of treatment. Historical records are permitted per investigator discretion.

1. Subject must have confirmation of non-acute promyelocytic leukemia (APL) Acute Myeloid Leukemia (AML) with a monocytic or monoblastic phenotype or a Ras pathway mutation. The subject's AML must be relapsed after or refractory to prior treatment with hypomethylating agent (HMA) and venetoclax combination.

   Note: other prior line(s) of therapy including stem cell transplant (SCT) are allowed, but HMA/Ven must be one of the preceding treatments. Subjects who have progressed to AML after prior treatment with HMA/Ven for high grade Chronic Myelomonocytic Leukemia (CMML) or Myelodysplastic Syndrome (MDS) are also eligible.
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
4. Adequate renal function as demonstrated by a calculated creatinine clearance ≥ 60 mL/min, calculated using the formula CKD-EPI Creatinine Equation (2021).
5. Adequate liver function, as demonstrated by:

   * Aspartate aminotransferase (AST) ≤ 3.0 x ULN*
   * Alanine aminotransferase (ALT) ≤ 3.0 x ULN*
   * Total bilirubin ≤ 1.5 x ULN, unless considered to be due to leukemic organ involvement or Gilbert's syndrome* *In subjects with Gilbert's syndrome, bilirubin needs to be ≤ 4 x ULN
6. Non-sterile male subjects must use contraceptive methods with partner(s) at least prior to beginning study drug administration and continuing up to 90 days after the last dose of study drug. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug. No contraception is required if male subjects are surgically sterile (vasectomy with medical assessment confirming surgical success) or if the male subject has a female partner who is postmenopausal or permanently sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
7. Female subjects must be either:

   * Postmenopausal: defined as age > 60 years with no menses for 12 or more months without an alternative medical cause; OR
   * Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy); OR
   * If subject is of childbearing potential, use of contraception is required while on study treatment and for 6 months after the last dose.
8. Subject must voluntarily sign an informed consent, approved by the Institutional Research Board (IRB), prior to the initiation of any research-related screening or study procedures.

Exclusion Criteria:

1. Subject has received prior treatment with cladribine for AML.
2. Subject has a white blood cell count > 25 x 109/L. Note: hydroxyurea and/or leukapheresis are permitted to meet this criterion.
3. Subject has known active central nervous system (CNS) involvement of AML.
4. Subject exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial, or fungal). Uncontrolled is defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment. Patients on antibiotics, antivirals, or antifungals with controlled systemic symptoms will not be excluded.
5. Subject has any clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study, including but not limited to:

   * New York Heart Association heart failure > class 2
   * Renal, neurologic, psychiatric, endocrine, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia.
6. Subject has a QTc interval > 470 msec.
7. Subject has a history of other malignancies within 2 years prior to study entry, with the following exceptions:

   * Adequately treated in situ carcinoma of the breast or cervix
   * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
   * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
   * Prostate cancer not requiring therapy beyond hormonal therapy
8. Subject is pregnant or breastfeeding.
9. Subject is known to be positive for HIV. HIV testing is not required.
10. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load. Hepatitis B or C testing is not required, and subjects with serologic evidence of prior vaccination to HBV may participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | End of Treatment, an average of 6 months
  Defined as the proportion of subjects who achieve a CR, CRi, or MLFS that is relapsed after or refractory to HMS/Ven

SECONDARY OUTCOMES:
Adverse Events | Duration of Treatment, an average of 6 months
  Frequency of adverse events (AEs) and serious adverse events (SAEs)
Event-free survival | Minimum of 3 years off study
  Event-free survival (EFS)
Overall survival | minimum of 3 years or off study
  Overall survival (OS)
Duration of response | minimum of 3 years or off study
  Duration of response (DOR)
Measurable residual disease | Baseline through End of Treatment, an average of 6 months
  Rate of measurable residual disease (MRD)-negativity

CONTACTS AND LOCATIONS:
Overall Officials: Christine McMahon, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universtiy of Colorado Hospital, Aurora, Colorado, United States